CLINICAL TRIAL: NCT06033755
Title: A Multidimensional Strategy to Managing Dysfunctional Breathing and Exercise-induced Laryngeal Obstruction in Adolescent Athletes
Brief Title: Managing Dysfunctional Breathing and Exercise-induced Laryngeal Obstruction in Adolescent Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VID Specialized University (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC 2016/1723
Record Dates: First submitted 2023-08-27; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Exercise Induced Laryngeal Obstruction (EILO)
Keywords: EILO; Physiotherapy intervention; Dysfunctional breathing; Adolescent athletes; Diaphragmatic breathing; Postural alignment

STUDY DESIGN:
Intervention Model Description: A mixed methods design, which combined qualitative and quantitative research, was used. Data, including subjective experiences of respiratory distress, findings from physiotherapeutic body examinations and objective measurements of lung function and aerobic capacity were gathered before and after a five month intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with EILO were recruited and given treatment (i.e. one arm?) (Other): Only participants with EILO were recruited and given treatment as usual.
  Interventions: Other: Norwegian psychomotor physiotherapy

INTERVENTIONS:
Other: Norwegian psychomotor physiotherapy — The intervention consisted predominantly of Norwegian Psychomotor Physiotherapy (NPMP) in which participants received individually tailored treatment based on the body examination and reported respiratory distress. NPMP addresses bodily tension, postural de-alignments and dysfunctional breathing patterns. The consultations also included a cognitive dimension, that is a conversation, in which thoughts and behaviours about training and competing were addressed and where participants were provided with "self help" measures that could improve breathing during training and competing. A rehabilitation plan for each participant was designed to limit further impairments and maintaining aerobic capacity without intensifying EILO symptoms. The intervention lasted 5 months.
  Other Names: Elements of cognitive behavioural therapy; Rehabilitation plan

SUMMARY:
This study aimed to assess if a multidimensional individually tailored intervention, including Norwegian Psychomotor Physiotherapy (NPMP), elements of cognitive behavioural therapy and a rehabilitation plan, helped reduce inspiratory distress and dysfunctional breathing in adolescent athletes with EILO. A mixed methods design, which combined qualitative and quantitative research, was used. Data, including subjective experiences of respiratory distress, findings from NPMP body examinations and objective measurements of lung function and aerobic capacity were gathered before and after a five month intervention involving 18 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent athletes with symptoms of EILO
* Referred to Norwegian Psychomotor Physiotherapy

Exclusion Criteria:

* Other respiratory symptoms
* Additional diagnosis

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Subjective experiences of respiratory distress associated with exercise reported descriptively in an interview pre and post treatment | Five months
  Experiences of respiratory distress were explored through a history taking and in an qualitative interview based on a questionnaire developed by O. Roksund (2012) Larynx in exercising humans - the unexplored bottleneck of the airways. University of Bergen Norway (PhD thesis). The questionnaire is not developed for research purposes, and reliability and validity studies are lacking. It is however, functional as a basis for the pre and post interview in which respiratory distress was explored and is commonly used for the same purpose at Haukeland University hospital in Norway. The reporting was descriptive and qualitative, and no scale or scores were used.

CONTACTS AND LOCATIONS:
Overall Officials: Liv-Jorunn Kolnes, PhD, Principal Investigator — VID Specialized University
Locations (1):
- Liv-Jorunn Kolnes, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The descriptive datasets concerning the body examinations generated during the study will not be publicly available du to individual privacy concerns, but will be available from the lead investigator on reasonable request.
Supporting Information: SAP
Time Frame: All statistical material will be published in the article depicting the study. This will be submitted during august/september 2023.

REFERENCES:
- [Derived] Kolnes LJ, Stensrud T, Andersen OK. A multidimensional strategy to managing dysfunctional breathing and exercise-induced laryngeal obstruction in adolescent athletes. BMC Sports Sci Med Rehabil. 2024 Jan 11;16(1):13. doi: 10.1186/s13102-023-00804-2. PMID 38212851